CLINICAL TRIAL: NCT01948414
Title: Cognitive Processes Study in Obese Women With and Without Eating Disorders : Research of Electro-physiological Similarity With Addiction
Brief Title: Cognitive Processes Study in Obese Women With and Without Eating Disorders
Acronym: P300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012.784
Record Dates: First submitted 2013-09-02; First posted 2013-09-23 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hyperalimentation and Obesity
Keywords: Obesity; Hyperalimentation; Event-Related Potential; P300
MeSH Terms: conditions — Hyperphagia; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- obese women with eating disorders (Other): Obese women with eating disorders : women with BMI higher or equal 35 and disinhibition score to TFEQ strictly higher to 8
  Interventions: Procedure: electroencephalography; Biological: Blood sampling; Behavioral: Questionnaires regarding eating habits (TFEQ, EDI) and anxiety/depression (HAD)
- Obese women without eating desorders (Other): Obese women without eating disorders : women with BMI higher or equal to 35 and disinhibition score to TFEQ lower or equal to 8
  Interventions: Procedure: electroencephalography; Biological: Blood sampling; Behavioral: Questionnaires regarding eating habits (TFEQ, EDI) and anxiety/depression (HAD)
- Lean women (Other): Lean women : women with BMI from 18.5 to 24.5 and disinhibition score to Three-Factor Eating Questionnaire (TFEQ)lower or equal to 8
  Interventions: Procedure: electroencephalography; Biological: Blood sampling; Behavioral: Questionnaires regarding eating habits (TFEQ, EDI) and anxiety/depression (HAD)

INTERVENTIONS:
Procedure: electroencephalography
Biological: Blood sampling
Behavioral: Questionnaires regarding eating habits (TFEQ, EDI) and anxiety/depression (HAD)

SUMMARY:
The P300 is one of the cognitive wave of the Event-Related Potential (ERP) that is used to investigate the cognitive process. The P300 component are accepted as electro-physiological markers of neuropsychiatric disorders like alcoholism or drug addiction.

Recent scientific data suggest that eating disorders, leading to weight gain and obesity, will be similar of those of drug addiction: it is the incentive sensitization theory that implicates the dopaminergic reward system.

The aim of this cross-sectional study is to investigate the alteration of P300 auditory ERP in obese women with eating disorders in comparison with obese and lean women without eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* women
* Aged from 20 to 55 years
* Fasting glycemia under 7mmol/L
* Lean women : women with BMI from 18.5 to 24.5 and disinhibition score to Three-Factor Eating Questionnaire (TFEQ)lower or equal to 8
* Obese women without eating disorders : women with BMI higher or equal to 35 and disinhibition score to TFEQ lower or equal to 8
* Obese women with eating disorders : women with BMI higher or equal 35 and disinhibition score to TFEQ strictly higher to 8

Exclusion Criteria:

* Subject not in compliance with the recommendations of French National Law in force
* Medical history of diabetes and surgery history of obesity
* Drug use that could affect the ERP recording
* Hospital Anxiety and Depression scale : evaluation subscale (anxiety and/or depression) strictly higher to 11

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
P300 amplitude | At the beginning of the exploration visit (when patient is fasting) that will take place between 1 and 15 days after inclusion
  The auditory event-related potentials measure will be elicited with an auditory oddball paradigm. The activity will be recorded thanks to electroencephalography from frontal, central and parietal electrodes, using an electrode cap.

SECONDARY OUTCOMES:
Auditory ERP ( latency P300, amplitude and latency of N2 wave recorded from frontal, central and parietal electrode) | fasting (up to 15 days)
  The technique of auditory ERP will be an auditory discriminated task paradigm
assessment of dietary restraints and disinhibition | fasting (up to 15 days)
  Participants will complete self-report questionnaires including Three-Factor Eating Questionnaire and Eating Disorders Inventory. The lean subjects should not have TFEQ disinhibition score more than 8. The obese subjects will be separated on two groups depending on TFEQ dishinibition score (strictly greater than 8, the obese with eating disorder, less than or equal 8, obese without eating disorder).
glucose, insulin, leptin and ghrelin plasmatic rate | fasting (up to 15 days)
  respectively reverse-phase high-performance liquid chromatography (RP-HPLC), ImmunoRadio Metric (IRMA) and ELISA assay
dopamine D2 receptor Taq 1 polymorphism | fasting (up to 15 days)
  Real time PCR
Dietary intake and eating patterns | At day 1 and at day 15
  Women will be interviewed by dietician, using a 24 h food questionnaire with additional questions regarding health and eating habits

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, Pratician, Principal Investigator — CRNH Rhône-Alpes /CENS Centre Européen pour la Nutrition et la Santé - Centre Hospitalier Lyon Sud
Locations (1):
- CRNH Rhône-Alpes /CENS Centre Européen pour la Nutrition et la Santé Centre Hospitalier Lyon Sud - Pavillon médical 165, chemin du Grand Revoyet, Pierre-Bénite, France

REFERENCES:
- [Result] Iceta S., Benoit J., Lambert-Porcheron S., Peyrat J., Cristini P., Poulet E., Laville M., Disse E. Obésité, addiction et prise alimentaire : étude des potentiels évoqués cognitifs. Nutrition Clinique et Métabolisme. 2018;32:231-338 (Section " 232 Congrès ", résumé CO09). doi:10.1016/j.nupar.2018.09.007 / 2018.09.008
- See also: Related Info — http://www.crnh-rhone-alpes.fr